CLINICAL TRIAL: NCT00167453
Title: Evaluation of the Benefits of a Group Exercise Program and a Group Exercise and Education Program for Individuals With Parkinson's Disease (BEEP)
Brief Title: Benefits of Exercise and Education for Individuals With Parkinson's Disease (BEEP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bio-REB 05-71
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2006-09

CONDITIONS: Parkinson Disease
Keywords: Nervous system disease; movement disorder; exercise; balance; education
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases; Movement Disorders; Motor Activity | interventions — Exercise; Educational Status

INTERVENTIONS:
Procedure: Exercise, Education

SUMMARY:
The research outlined in the BEEP proposal aims to test whether a 12 week exercise program alone or combined with a 12 session education program will benefit the physical, emotional and social well being of individuals in early to mid stages of Parkinson's Disease compared to a Control group and whether these benefits are maintained once the programs are complete and over the following 9 months.

DETAILED DESCRIPTION:
The BEEP proposal tests whether a 12 week exercise program alone or combined with a 12 session education program will benefit the physical, emotional and social well being of individuals in early to mid stages of Parkinson's Disease and whether these benefits are maintained once the programs are complete.

This is a single blind randomized control trial with pretest and posttests after a 3 month intervention and subsequent follow-up testing at 3 months and 9 months post intervention. The Intervention groups (group exercise, group exercise and education) will be compared to a control group and to each other. Each group will have 15 participants.

The study compares the interventions and control groups to determine the following health outcomes:

* physical performance
* levels of physical and social activity
* perceived quality of life
* perceived self efficacy for managing chronic neurological disease

Analysis of variance will be used to test for group differences.

The Interventions: Exercise Group: Two, 75 minute sessions per week for 24 sessions. Program components include flexibility and strengthening exercises, balance and posture training, practice of functional tasks and endurance training. Education and Exercise Group: Exercise, same as for Exercise Group, delivered simultaneously to both intervention groups.

Education: One, 75 minute session per week for 12 sessions at RUH, including:

* disease process and clinical presentation
* medication use in PD
* benefits of exercise
* managing movement difficulties and tips for performance of functional activities
* assistive devices for improved independence and safety
* driving
* prevention of falls: movement strategies and home modifications to increase safety
* speech, swallowing and facial expression
* nutrition and weight maintenance, managing constipation
* managing changes in mood & emotions, managing personal relationships
* coping with life changes caused by PD
* relaxation methods

Monitoring will occur to limit "informal" education that might occur during the exercise program from this group to the pure Exercise Group.

Control Group: no intervention The proposed study will add to the body of evidence evaluating the immediate and longer term benefits of group exercise programs for individuals with PD and will evaluate the benefits gained by adding an education program to an exercise program intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease or Parkinson Syndrome
* Stages I-III of disease progression
* Between 40 and 80 years of age

Exclusion criteria:

* Acute illness
* History of significant cardio-pulmonary insufficiency/illness or any other condition which limits physical activity.
* History of neurological disorder other than Parkinson Disease
* Diagnosis of dementia or significant cognitive impairments.
* Mental State Exam (Folstein et al, 1975) score of < 20
* Beck Depression Inventory-II score of > 20 will be excluded.
* Participation in an organized community exercise program in the past 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2005-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
all variables measured at baseline, post intervention, months following, and 9 months following.
Stanford Self-Efficacy for Managing Chronic Disease
The Activities-specific Balance Confidence (ABC) Scale
Timed Up and Go Test(TUG)

SECONDARY OUTCOMES:
Northwestern University Disability Scale:
Schwab & England ADL Scale:) independence in ADL
Parkinson's Disease Questionnaire - Short Form (PDQ - 8):
Beliefs about Symptom Specific Expectancies:
Social and Physical Activities Questionnaire:

CONTACTS AND LOCATIONS:
Overall Officials: M Suzanne Sheppard, PhD, Principal Investigator — Saskatoon Health Region
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886